CLINICAL TRIAL: NCT01597648
Title: A Randomized, Open-Label, Crossover Study to Evaluate the Bioequivalence of a Combined Formulated Tablet Compared With Maraviroc and Combivir™ Administered Concurrently in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Bioequivalence of a Combined Formulated Tablet Compared With Maraviroc and Combivir™
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 115325
Record Dates: First submitted 2012-05-03; First posted 2012-05-14 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: Combivir™, HIV, bioequivalence, Combined Formulated Tablet, Combined Formulated Tablet, HIV, bioequivalence, Combivir, Selzentry™, Celsentri™, lamivudine, zidov
MeSH Terms: conditions — Infections | interventions — Maraviroc; lamivudine, zidovudine drug combination

ARMS (2):
- Sequence 1 (Experimental): Treatment A: 1 tablet of GSK2838510 (maraviroc 300 mg, lamivudine 150 mg, and zidovudine 300 mg as a combined formulation) after an overnight fast Washout Treatment B: 1 tablet of maraviroc 300 mg + 1 tablet of Combivir taken concurrently after an overnight fast.
  Interventions: Drug: Maraviroc; Drug: Combivir; Drug: GSK2838510
- Sequence 2 (Experimental): Treatment B: 1 tablet of maraviroc 300 mg + 1 tablet of Combivir taken concurrently after an overnight fast.
  Washout Treatment A: 1 tablet of GSK2838510 (maraviroc 300 mg, lamivudine 150 mg, and zidovudine 300 mg as a combined formulation) after an overnight fast
  Interventions: Drug: Combivir

INTERVENTIONS:
Drug: Maraviroc — 300 mg
  Arms: Sequence 1
Drug: Combivir — 1 tablet: lamivudine 150mg, zidovudine 300mg
Drug: GSK2838510 — Maraviroc 300mg, lamivudine 150mg, zidovudine 300mg
  Arms: Sequence 1

SUMMARY:
This is a study in healthy adult subjects to evaluate the bioequivalence of a Combined Formulated Tablet compared with maraviroc and Combivir administered concurrently versus maraviroc + Combivir. 42 subjects will be enrolled in the study such that 40 subjects complete dosing and critical assessments. The total duration of a subject's participation will be approximately 33 to 35 days, including a screening period (Day -21 to Day -1), 2 treatment periods (Days 1-3), at least a 7-day washout between Period 1 and Period 2, and a follow-up visit 7 to 14 days after the last dose of study drug in Period 2. Each dosing period will begin the evening prior to dosing and extend until 48 hours (Day 3) after dosing. Subjects will be randomly assigned to receive 1 of the following 2 treatments in Period 1 then crossover to receive the alternate treatment in Period 2:

In Sequence 1 (N=21) subjects will receive Treatment A followed by a 7 day washout and Treatment B. In Sequence 2 (N=21) subjects will receive Treatment B followed by a 7 day washout and Treatment A. Treatment A consists of 1 tablet of maraviroc 300 mg, lamivudine 150 mg, and zidovudine 300 mg as a combined formulation after an overnight fast. Treatment B consists of 1 tablet of maraviroc 300 mg + 1 tablet of Combivir taken concurrently after an overnight fast. On Day 1 of each treatment period, subjects will receive study drug in the morning after an overnight fast of at least 8 hours. Study drug will be administered with 240 mL of water. Dosing in each treatment period will be separated by a minimum washout period of at least 7 days between doses. All subjects will undergo safety and other assessments. Subjects may be discharged after all study procedures are completed on the morning of Day 3, with instructions to return for the next study period or the follow-up visit, as appropriate. The follow-up visit will occur 7 to 14 days after the last dose of study drug in Period 2. Pharmacokinetic blood samples will be collected during each treatment period for evaluation of maraviroc, lamivudine, and zidovudine before dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, and 48 hours after dosing (total of 16 PK time points per treatment period). Protocol waivers or exemptions are not allowed, with the exception of immediate safety concerns. Therefore, adherence to the study protocol requirements, including those specified in the Time and Events Table, are essential and required for study conduct.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to 55 years of age (inclusive); healthy as determined by a responsible physician, based on a medical evaluation, including medical history, vital sign measurements, physical examination, clinical laboratory tests, and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A female subject is eligible to participate if she is of: Non childbearing potential, defined as premenopausal females with a documented tubal ligation or hysterectomy; or postmenopausal, defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle stimulating hormone [FSH] greater than 40 MlU/mL and estradiol less than 40 pg/mL (less than 146.8 pmol/L) is confirmatory). Childbearing potential and is abstinent (abstinence from penile-vaginal intercourse must be consistent with the preferred and usual lifestyle of the subject) or agrees to use 1 of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 30 days after the study.
* The subject has alanine aminotransferase, alkaline phosphatase, and bilirubin less than and equal to 1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is less than 35%).
* Subject has a QTcB <450 msec.
* The subject has a body mass index (BMI) between 18.5 and 31.0 kg/m2 (inclusive) and a total body weight greater than and equal to 45 kg for females and ≥50 kg for males.
* The subject provides written informed consent.
* The subject is a current nonsmoker greater than 3 months.

Exclusion Criteria:

* The subject has a positive prestudy drug/alcohol screen. At minimum, the drug screen will include alcohol, cotinine, amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* The subject has a history of sensitivity to any of the study drugs, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates the subject's participation.
* The subject is unable to refrain from the use of prescription or nonprescription drugs, including vitamins and herbal and dietary supplements (including St. John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug, unless in the opinion of the investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has a history of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 14 drinks/week for men or greater than 7 drinks/week for women.
* The subject has consumed red wine, Seville oranges, grapefruit, or grapefruit juice within 7 days prior of the first dose of study drug.
* The female subject is pregnant as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or before dosing.
* The female subject is lactating.
* The subject is unwilling or unable to follow the procedures outlined in the protocol.
* The subject has a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic, and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study drugs. A subject with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease, or pancreatitis should be excluded.
* The subject has a positive prestudy hepatitis B surface antigen, hepatitis C antibody, or HIV antibody result.
* The subject has a history of Gilbert's disease.
* The subject's participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* The subject has systolic blood pressure outside the range of 90-140 mmHg, diastolic blood pressure outside the range of 45-90 mmHg, or heart rate outside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects. A single repeat measurement is allowed for eligibility determination.
* The subject meets any of the following exclusion criteria for the screening ECG (a single repeat ECG is allowed for eligibility determination): Males heart rate: less than 45 or greater than 100 bpm; females heart rate: less than 50 or greater than 100 bpm; Males and females PR interval: less than 120 or greater than 220 msec; Males and females QRS duration: less than 70 or greater than 120 msec; Males and females QTcB: greater than 450 msec. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [2nd degree or higher], and Wolf Parkinson White syndrome). Sinus pauses greater than 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and Medical Monitor, will interfere with the safety for the individual subject. Nonsustained or sustained ventricular tachycardia (greater than and equal to 3 consecutive ventricular ectopic beats).
* The subject is unwilling or unable to follow the procedures outlined in the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety parameters: AEs, vital signs, ECG, body temperature and laboratory assessments, including haematology, clinical biochemistry and cardiac troponin | Approximately 5 weeks from first dose to the follow-up visit
  To assess the safety and tolerability of single and repeat inhaled doses of GSK2339345 administered by an aqueous droplet inhaler
Assessment of oropharyngeal sensation perturbation via a 4 point scale | Approximately 5 weeks from first dose to the follow-up visit
  To assess the changes in oropharyngeal sensation caused by single and repeat inhaled doses of GSK2339345 administered by an aqueous droplet inhaler

SECONDARY OUTCOMES:
Plasma concentrations of GSK2339345 and single and repeat dose derived pharmacokinetic parameters including Cmax, tmax, AUC(0-t), AUC(0-inf), and AUC(0- τ), as appropriate where data allow | Approximately 5 weeks from first dose to the follow-up visit
  To evaluate the systemic pharmacokinetics of single and repeat doses of inhaled GSK2339345 in healthy volunteers administered by an aqueous droplet inhaler
Identification of taste of the solution and rating on 11 point scale to rate pleasantness or unpleasantness | Approximately 5 weeks from first dose to the follow-up visit
  To assess the palatability of GSK2339345 administered by an aqueous droplet inhaler

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline